CLINICAL TRIAL: NCT03690648
Title: Genetic Factors and Immunological Determinism of Persistent Consequences of Chikungunya Fever: Genome-wide Association Study
Brief Title: Genetic Factors and Immunological Determinism of Persistent Consequences of Chikungunya
Acronym: CHIKGENE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Collaborators: Conservatoire national des Arts et Métiers (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/CHU/12
Record Dates: First submitted 2018-09-26; First posted 2018-10-01 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Chikungunya Fever
MeSH Terms: conditions — Chikungunya Fever | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva and blood collection for genetical analysis (GWAS)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Saliva collection: * Clinical examination;
  * Quality of life survey;
  * Saliva collection for genetical analysis
  Interventions: Other: Quality of life survey; Genetic: Saliva collection
- Saliva and Blood collection: * Clinical examination;
  * Quality of life survey;
  * Saliva and blood collection for genetical analysis
  Interventions: Other: Quality of life survey; Genetic: Saliva collection; Genetic: Blood collection

INTERVENTIONS:
Other: Quality of life survey — Administration of scales: SF-12v2, EQ-5D, QCD, DN4, EIMIR, MFIS-5 et EHAD
Genetic: Saliva collection — Collection of 20 ml of saliva with a kit of saliva collection
Genetic: Blood collection — Collection of 20 ml of blood with kit of blood collection
  Groups: Saliva and Blood collection

SUMMARY:
Chikungunya virus (CHIKV) infection has become a threat to public health worldwide. Reunion Island, due to the 2005-2006 epidemic, has acquired unique expertise and remains at the forefront of global research on this disease. The idea of genetic determinism of the clinical expression of infectious diseases has been supported by many epidemiological arguments over the past fifty years. The identification of genetic variants, associated with a disease, often allows a better understanding of the molecular mechanisms involved with consequent significant benefits such as the development of specific biomarkers for new preventive (vaccination) and / or therapeutic (drug design) approaches. In the absence of well-documented hypotheses about the genes potentially involved in the occurrence or evolution of a disease, genome-wide association studies (GWAS), whole genome, of nucleotide polymorphisms (SNPs) and the principle of linkage disequilibrium, under the commonly accepted hypothesis that the expression of a common disease is based on a small number of alleles commonly found in the population (frequency of minor allele greater than 1-5%), have become a method of choice, free of hypothesis, to specify the part of heritability of a complex disease and to identify its genetic determinants. Several epidemiological arguments support a significant proportion of genetic determinism in the explanation of the evolutionary pattern of Chikungunya, whose proportion of chronic forms can reach 40-60% in population-based studies conducted in the two years following an epidemic:

* There are few risk factors associated with chronic forms and these appear to be unclear (age, comorbidities with several elements of the metabolic syndrome) or inconsistent (immune burden) in population studies;
* The incidence of severe or atypical forms is rare in the order of 1% of infections;
* In contrast to the acute phase (J1-J21) for which there seems to be a role of the viral load intensity and a consensual pro-inflammatory immune signature according to a recent meta-analysis]; The role of the intensity of the viral load in the pathogenesis of chronic arthralgia (> J90) and their immune signature remain to be determined, the latter being rather nonspecific, according to studies conducted in Reunion, Italy or Singapore.

These elements justify the interest of a GWAS in the Chikungunya to identify new avenues and mechanistic hypotheses likely to explain the chronic arthralgia characteristic of the disease.

ELIGIBILITY:
Inclusion Criteria:

* -Subject of the seroprevalence survey or neighbor living in the same neighborhood likely to confirm an exposure status or known;
* Exposure status established by specific IgG serology, collected between March 1st, 2005 and December 31st, 2006;
* Affiliated to a social security scheme;
* Age between 18 and 75 years old;
* Paternal and maternal 1st and 2nd degree ascendants (parents and grandparents) and at least 3 generations of the family present on the island (grandparents born on the island of Réunion);
* Able to spit

Exclusion Criteria:

* Exposure status unknown;
* Absence of social security;
* Age <18 years and> 75 years;
* Physical inability to spit;
* Pregnant women;
* Protected person (tutorship or curatorship).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject with a serological status known for Chikungunya virus for the period between March 1st, 2005 and December 31st, 2006 (epidemic period in reunion Island).
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
identify by a genome-wide association study the genetic factors associated with the evolutionary profile of Chikungunya | through study completion, an average of 1 year
  to determine if certain genetic profiles may be predictive of progression to asymptomatic or acute disease, or to the chronic character of the manifestations of the disease

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de La Réunion, Saint-Pierre, Reunion

IPD SHARING:
Plan to Share IPD: No